CLINICAL TRIAL: NCT03512028
Title: Effects of Remote Limb Ischemic Conditioning to Enhance Performance, Cognitive-motor Learning and Muscle Strength in Healthy Young Adults
Brief Title: Remote Limb Ischemic Conditioning to Enhance Learning and Muscle Strength in Healthy Young Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Catherine E. Lang, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIHR01HD085930-Aim1; R01HD085930 (NIH)
Record Dates: First submitted 2018-04-16; First posted 2018-04-30 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Healthy, Young Adults
Keywords: ischemic conditioning, motor learning, strength, cognition

STUDY DESIGN:
Intervention Model Description: Single blinded, randomized controlled trial
Who Masked: Participant
Masking Description: Participants are masked to group assignment (RLIC vs. Sham conditioning).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Limb Ischemic Conditioning (RLIC) (Experimental): RLIC is achieved via blood pressure cuff inflation to 20 mmHg above systolic blood pressure on the dominant arm. RLIC requires 45 minutes and involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. RLIC is performed on visits 1-8.
  Interventions: Behavioral: RLIC; Behavioral: Muscle strength training; Behavioral: Driving training; Behavioral: Balance training
- Sham Conditioning (Sham Comparator): Sham conditioning is achieved via blood pressure cuff inflation to 10 mmHg under diastolic blood pressure on the dominant arm. Sham conditioning requires 45 minutes and involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. Sham conditioning is performed on visits 1-8.
  Interventions: Behavioral: Sham conditioning; Behavioral: Muscle strength training; Behavioral: Driving training; Behavioral: Balance training

INTERVENTIONS:
Behavioral: RLIC — See descriptions under arm/group descriptions. RLIC is delivered for 8 visits. Visits 1-3 occur on consecutive work days and visits 4-8 occur on alternating week days.
  Other Names: remote limb ischemic conditioning
  Arms: Remote Limb Ischemic Conditioning (RLIC)
Behavioral: Sham conditioning — See descriptions under arm/group descriptions. Sham conditioning is delivered for 8 visits. Visits 1-3 occur on consecutive work days and visits 4-8 occur on alternating week days.
  Arms: Sham Conditioning
Behavioral: Muscle strength training — All participants undergo muscle strength training of the wrist extensor muscles on one side. Strength training follows standard American College of Sports Medicine guidelines for frequency, intensity, progression etc. Strength training is provided at visits 3-8
Behavioral: Driving training — All participants undergo training of a complex cognitive-motor task using a driving simulator. Participants learn to 'drive' on a virtual course, maximizing speed and minimizing errors. Participants perform the driving task once each day for visits 3-8.
Behavioral: Balance training — All participants undergo training on a balance board, learning to hold the board level with equal weight on each leg. Participants perform the balance task for 15, 30-second trials per day at visits 3-8.

SUMMARY:
The purpose of this research study is to determine if remote limb ischemic conditioning (RLIC) can enhance learning of a motor (balance) and an ecologically valid, complex cognitive-motor (driving) task, and increase skeletal muscle strength in neurologically-intact young adults.

DETAILED DESCRIPTION:
Ischemic conditioning is an endogenous phenomenon in which exposing a target organ or tissue to one or more brief episodes of ischemia results in protection of that organ against subsequent ischemia. The effects of ischemic conditioning are not confined within an organ but can be can be transferred from one organ to another, a technique called remote ischemic conditioning. A clinically feasible method for this is remote limb ischemic conditioning (RLIC), where episodes of ischemia and perfusion are induced with a blood pressure cuff placed on the arm.

The overall goal of this line of work is to use ischemic conditioning to enhance learning and outcomes in persons with neurologic injuries. Two previous studies have shown that remote limb ischemic conditioning (RLIC) can enhance learning a motor task in healthy young adults. The current study extends that work to determine if RLIC enhances muscle strength training and a complex cognitive-motor task (simulated driving). This Phase I study will yield the necessary information to design and execute subsequent trials in neurologic patient populations.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between the age of 18 and 40 years
2. Visual acuity of 20/20 with corrected vision

Exclusion Criteria:

1. History of neurological condition (i.e. stroke, Alzheimer's disease, Parkinson's disease), Attention Deficit Hyperactivity Disorder (ADHD), depression, bipolar disorder, balance impairment, or vestibular disorder
2. History of severe motion sickness, moderate to severe motion sickness or nausea on oculo-motor components of Simulator sickness questionnaire, inability to ride a car, boat, train or airplane due to motion sickness
3. Recent wrist, hand or forearm injury that would currently prevent ability to lift weights
4. History of lower extremity condition, injury, or surgery that would currently impair ability to stand or balance
5. Any extremity soft tissue, orthopedic, or vascular injury (i.e. peripheral vascular disease) which may contraindicate RLIC
6. Any cognitive, sensory, or communication problem that would prevent completion of the study
7. History of or current sleep apnea
8. Current intensive weight lifting or interval training exercise
9. Current substance abuse or dependence
10. Unwillingness to travel for all study visits

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, all of the individual participant data after deidentification will be submitted to Washington University data repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication of results. No ending date
Access Criteria: Data will be available to anyone who wishes to access it through Washington University data repository.
URL: https://openscholarship.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Remote Limb Ischemic Conditioning (RLIC): RLIC is achieved via blood pressure cuff inflation to 20 mmHg above systolic blood pressure on the dominant arm. RLIC requires 45 minutes and involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. RLIC is performed on visits 1-8.
  RLIC is delivered for 8 visits. Visits 1-3 occur on consecutive work days and visits 4-8 occur on alternating week days.
  Muscle strength training: All participants undergo muscle strength training of the wrist extensor muscles on one side. Strength training follows standard American College of Sports Medicine guidelines for frequency, intensity, progression etc. Strength training is provided at visits 3-8
- Sham Conditioning: Sham conditioning is achieved via blood pressure cuff inflation to 10 mmHg under diastolic blood pressure on the dominant arm. Sham conditioning requires 45 minutes and involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation. Sham conditioning is performed on visits 1-8.
  Sham conditioning is delivered for 8 visits. Visits 1-3 occur on consecutive work days and visits 4-8 occur on alternating week days.
  Muscle strength training: All participants undergo muscle strength training of the wrist extensor muscles on one side. Strength training follows standard American College of Sports Medicine guidelines for frequency, intensity, progression etc. Strength training is provided at visits 3-8
Period: Overall Study
Arm/Group | Remote Limb Ischemic Conditioning (RLIC) | Sham Conditioning
Started | 19 | 15
Completed | 15 | 15
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remote Limb Ischemic Conditioning (RLIC) | Sham Conditioning | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (3.8) | 27.3 (4.3) | 26.4 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 8 | 8 | 16
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
BMI [Mean (Standard Deviation); unit: kg/m*m] | 22.6 (3.1) | 24.6 (3.9) | 23.6 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: One-repetition Maximum of Wrist Extensors
Description: The maximum amount of force (lbs) that a participant can generate while performing one wrist extension movement.
Time Frame: Pre-intervention, post-intervention (2 weeks later), and 1 month post-intervention follow-up
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Remote Limb Ischemic Conditioning (RLIC) | Sham Conditioning
Number analyzed (Participants) | 15 | 15
lbs
  Pre | 22.6 (10.3) | 23.7 (7.9)
  Post | 32.0 (14.0) | 29.9 (10.8)
  Follow-up | 30.8 (13.4) | 29.2 (10.5)
Statistical Analysis 1: Comparison: Remote Limb Ischemic Conditioning (RLIC) vs Sham Conditioning; Mixed model ANOVA with group (RLIC, Sham) and time (pre-, post-, and follow-up ). The main analysis of interest is the group x time interaction from pre- to post-; Test type: Superiority; p = 0.002, ANOVA — Interaction effect of group x time from pre- to post- intervention; Mean Difference (Net) = 3.2 — Estimated difference between slopes
Statistical Analysis 2: Comparison: Remote Limb Ischemic Conditioning (RLIC) vs Sham Conditioning; Test type: Superiority; p = 0.001, ANOVA — Main effect of time
Statistical Analysis 3: Comparison: Remote Limb Ischemic Conditioning (RLIC) vs Sham Conditioning; Test type: Superiority; p = 0.844, ANOVA — Main effect of group

ADVERSE EVENTS:
Time Frame: Duration of the intervention, which was two weeks.
Arm/Group | Remote Limb Ischemic Conditioning (RLIC) | Sham Conditioning
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 0/19 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT03512028/Prot_SAP_000.pdf